CLINICAL TRIAL: NCT05740995
Title: A Single-center, Prospective Cohort Study of Neoadjuvant Anti-PD-1 Plus Chemotherapy in Locally Advanced Resectable Esophageal Squamous Cell Carcinoma
Brief Title: Neoadjuvant Anti-PD-1 Plus Chemotherapy in Locally Advanced Resectable Esophageal Squamous Cell Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B2021-129
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Esophageal Squamous Cell Carcinoma; Neoadjuvant Chemoimmunotherapy
Keywords: Esophageal Squamous Cell Carcinoma; Neoadjuvant Chemoimmunotherapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Fresh biopsy and surgical specimen
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neoadjuvant Anti-PD-1 Plus Chemotherapy Group: Patients with locally advanced resectable ESCC (cT3-4aN0-1M0) who receive neoadjuvant anti-PD-1 plus chemotherapy and donate biological samples
  Interventions: Drug: neoadjuvant anti-PD-1 plus chemotherapy

INTERVENTIONS:
Drug: neoadjuvant anti-PD-1 plus chemotherapy — Patients will be given preoperative treatment as below once recruited:
  1. Chemotherapy is delivered and composed of two cycles of Nab-paclitaxel 135mg per square meter of body-surface area and cisplatin 75mg per square meter of body-surface area every 3 weeks;
  2. PD-1 antibody is delivered 200 mg (iv, in 30 minutes) every 3 weeks;
  3. After neoadjuvant therapy of 3-4 cycles, esophagectomy is performed. We advise starting 4 cycles of identical chemoimmunotherapy in 6w after surgery.

SUMMARY:
The purpose of this study is to evaluate the outcomes and identify predictors of neoadjuvant anti-PD-1 plus chemotherapy in locally advanced resectable esophageal squamous cell carcinoma (ESCC). In this single-center cohort study, we are aiming to (1) evaluate the therapeutic efficacy and survival benefits on patients with locally advanced resectable ESCC (cT3-4aN0-1M0); (2) evaluate the value of genomic indicators including MMR alternation status in predicting therapeutic responses and prognosis; (3) evaluate the value of transcriptomic indicators including B cell lineage features in predicting therapeutic responses and prognosis; (4) evaluate the value of microbial and metabolite indicators in predicting therapeutic responses and prognosis. Whole exome sequencing, RNA sequencing, 16S rRNA sequencing and Liquid Chromatography with tandem mass spectrometry (LC-MS-MS) of samples of patients to neoadjuvant chemoimmunotherapy before and after treatment are performed to explore the mechanisms of drug resistance and identification of predictive and prognosis biomarkers.

DETAILED DESCRIPTION:
Multiple clinical trials investigated the safety and feasibility of neoadjuvant anti-PD-1 plus chemotherapy in esophageal squamous cell carcinoma (ESCC). However, the efficacy of neoadjuvant chemoimmunotherapy was undetermined and existing biomarkers failed to provide stable prediction of therapeutic responses. This study seek to further evaluate the clinical outcomes and identify biological predictors of neoadjuvant anti-PD-1 plus chemotherapy in locally advanced resectable esophageal squamous cell carcinoma (ESCC). In this single-center cohort study, our aims include:

1. evaluate the therapeutic efficacy and survival benefits on patients with locally advanced resectable ESCC (cT3-4aN0-1M0);
2. evaluate the value of genomic indicators in predicting therapeutic responses and prognosis;
3. evaluate the value of transcriptomic indicators in predicting therapeutic responses and prognosis;
4. evaluate the value of microbial and metabolite indicators in predicting therapeutic responses and prognosis. Whole exome sequencing, RNA sequencing, 16S rRNA sequencing and Liquid Chromatography with tandem mass spectrometry (LC-MS-MS) of samples of responders and non-responders to neoadjuvant chemoimmunotherapy before and after treatment are performed to explore the mechanisms of drug resistance and identification of predictive and prognosis biomarkers, providing guidance to clinical decisions.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-confirmed squamous cell carcinoma of the esophagus;
2. Tumors of the esophagus are located in the thoracic cavity;
3. Pre-treatment stage as cT3-4aN0-1M0 (AJCC/UICC 7th Edition) (In case of stage cT4a, curative resectability has to be explicitly verified by the local surgical investigator prior to randomization).
4. Age is between 18 years and 75 years,
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-1;
6. Adequate cardiac function. All patients should perform ECG, and those with a cardiac history or ECG abnormality should perform echocardiography with the left ventricular ejection fraction > 50 %;
7. Adequate respiratory function with FEV1≥1.2L, FEV1%≥50% and DLCO≥50% shown in pulmonary function tests;
8. Adequate bone marrow function (White Blood Cells >4x10^9 /L; Neutrophil >2.0×10^9 /L; Hemoglobin > 90 g/L; platelets>100x10^9 /L);
9. Adequate liver function (Total bilirubin <1.5x Upper Level of Normal (ULN); Aspartate transaminase(AST) and Alanine transaminase (ALT)<1.5x ULN);
10. Adequate renal function (Glomerular filtration rate (CCr) >60 ml/min; serum creatinine (SCr) ≤120 µmol/L);
11. The patient has provided written informed consent and is able to understand and comply with the study;

Exclusion Criteria:

1. Patients with non-squamous cell carcinoma histology;
2. Patients with advanced inoperable or metastatic esophageal cancer;
3. Pre-treatment stage as cT1-2N0-1M0 (AJCC/UICC 7th Edition);
4. Pre-treatment stage as cN2-3 or cT4b(non-curatively-resectable verified by the local surgical investigator, AJCC/UICC 7th Edition);
5. Patients with another previous or current malignant disease which is likely to interfere with treatment or the assessment of response in the judgement of the local surgical investigator.
6. Any patient with a significant medical condition which is thought unlikely to tolerate the therapies. Such as cardiac disease (e.g. symptomatic coronary artery disease or myocardial infarction within last 12 months), clinically-significant lung disease, clinically-significant bone marrow, liver, renal function disorder;
7. Pregnant or lactating women and fertile women who will not be using contraception during the trial;
8. Allergy to any drugs;
9. Participation in another intervention clinical trial with interference to the therapeutic intervention during this study or during the last 30 days prior to informed consent;
10. Expected lack of compliance with the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced resectable ESCC (cT3-4aN0-1M0)
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Major pathological regression (MPR) rate | Up to the date of pathological reports obtained since the date of enrollment, up to 6 months
  The resected specimen following neo-adjuvant treatment are assessed by using standardised work up of the resection specimen in the pathology department and standardised histological criteria for tumour regression grading. MPR was defined as ≤10% residual viable tumor.

SECONDARY OUTCOMES:
Pathological response rate(pCR) | Up to the date of pathological reports obtained since the date of enrollment, up to 6 months
  The resected specimen following neo-adjuvant treatment are assessed by using standardised work up of the resection specimen in the pathology department and standardised histological criteria for tumour regression grading. PCR was defined as no evidence of vital residual tumor cells.
objective response rate (ORR) | 36 months after the last subject participating in
  ORR is evaluated by chest, abdominal & pelvic CT/MRI based on RESIST 1.1. Evaluation will be conducted every 6 weeks during neoadjuvant therapy and every 6 months after surgery.
overall survival (OS) | 36 months after the last subject participating in
  OS is defined as time interval from recruitment to all-caused death or censoring.
Progression-free survival(PFS) | 36 months after the last subject participating in
  Disease recurrence is defined as locoregional (esophageal bed or anastomotic or regional lymph nodes) or metastatic (supraclavicular lymph nodes or distant organs).
The correlation between detection of genomic, immune, microbial and metabolite features and the rate of therapeutic responses. | 36 months after the last subject participating in
  The detection of genomic, immune, microbial and metabolite features from biological samples before and after neoadjuvant chemoimmunotherapy is performed to analyze the correlation to treatment vulnerability.

CONTACTS AND LOCATIONS:
Overall Officials: Di Ge, MD, Study Director — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
The IPD will not be shared with other researchers in order to protect patients' privacy.